CLINICAL TRIAL: NCT03283748
Title: Detection of Motor Seizures Using Wireless Body Area Network
Brief Title: Detection of Motor Seizures Using WBAN
Acronym: DMS-WBAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mohawk College (Other)
Collaborators: Hamilton Health Sciences Corporation (Other); Toronto Metropolitan University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 3596
Record Dates: First submitted 2017-09-08; First posted 2017-09-14 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2018-03

CONDITIONS: Seizures, Tonic-Clonic
MeSH Terms: conditions — Seizures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Measurement of Motor Movements (Experimental): Wearable Accelerometer Sensors manufactured by leading manufacturers will be given to the participants to be worn around hands and legs. These sensors will be used to measure accelerations which will be impacted by the motor movements.
  Interventions: Device: Wearable sensors

INTERVENTIONS:
Device: Wearable sensors — Wearable sensors will be given to the participants to be worn and movement data will be collected

SUMMARY:
This study aims to collect the motor movement data using sensors to detect Generalized Tonic Clonic Seizures . Wearable sensors similar to smart watches will be used to detect seizures. The proposed system will consist of 3-4 wearable wireless sensor worn on the hands and legs. The data from these sensors will be send to the clod and collected to a central hub for analysis and detection of GTC Seizures.

DETAILED DESCRIPTION:
The key of the project is digital signal processing of the movement data collected. The medical application sensors from Analog Devices will be worn around the wrist and legs of the participants. These sensors will continuously collect the motor movement data. The data will be send to the cloud from where it will be collected at a central hub for digital signal processing and detection. The data analysis results will be compared with the standard EEG results for Tonic Clonic seizures and results will be verified.

ELIGIBILITY:
Inclusion Criteria:

* subject has seizures or symptoms of seizures

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-02-25 (Actual); Study Completion 2019-01-30 (Actual)

PRIMARY OUTCOMES:
Measurement of Acceleration | 3 months
  Motor movements will cause changes in acceleration. Accelerometer sensors will be used to measure the acceleration as a first step towards detection of Tonic Clonic Seizures

SECONDARY OUTCOMES:
Digital Signal processing of the data | 3 months
  The raw acceleration data collected will be processed in a computer with MATLAB software using Digital Signal processing techniques. These techniques will help identify the data and differentiate the seizure movements from normal movements thereby helping to detect seizures data

CONTACTS AND LOCATIONS:
Overall Officials: Mini Thomas, M.Eng., Principal Investigator — Mohawk College
Locations (1):
- Mini Thomas, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Non-EEG based ambulatory seizure detection designed for home use: What is available and how will it influence epilepsy care? — https://www.ncbi.nlm.nih.gov/pubmed/26926071
- See also: Detection of generalized tonic-clonic seizures by a wireless wrist accelerometer: A prospective, multicenter study — https://www.researchgate.net/publication/235520022_Detection_of_generalized_tonicclonic_seizures_by_a_wireless_wrist_accelerometer_A_prospective_multicenter_study
- See also: Electromyography-based seizure detector: Preliminary results comparing a generalized tonic-clonic seizure detection algorithm to video-EEG recordings — https://www.ncbi.nlm.nih.gov/pubmed/26190150
- See also: Safe and sound? A systematic literature review of seizure detection methods for personal useSafe and sound? A systematic literature review of seizure detection methods for personal use — https://www.ncbi.nlm.nih.gov/pubmed/26859097